CLINICAL TRIAL: NCT04006041
Title: A Phase II Trial of Combination of Toripalimab and Neoadjuvant Chemoradiotherapy in Esophageal Squamous Cell Carcinoma
Brief Title: Combination of Toripalimab and Neoadjuvant Chemoradiotherapy in Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jianhua Fu (Other)
Responsible Party: Sponsor-Investigator, Jianhua Fu, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TORINEOEC
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Esophageal Squamous Cell Carcinoma by AJCC V8 Stage; Resectable Esophageal Cancer
Keywords: Esophageal squamous cell carcinoma; Neoadjuvant chemoradiotherapy; Toripalimab; Pathologic complete response
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Pathologic Complete Response | interventions — toripalimab; TP protocol; Radiotherapy, Intensity-Modulated; Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab group (Experimental): All patients will receive standard fractionation radiation therapy (RT) scheme: 44Gy in 20 fractions over 4 weeks, concurrently with 4 cycles of paclitaxel/cisplatin (paclitaxel 50mg/m2 and cisplatin 25 mg/m2) on days 1, 8, 15, 22 and 2 cycles of toripalimab 240 mg on days 1, 22. Esophagectomy is performed 6-8 weeks after CRT completion.
  Interventions: Drug: Toripalimab; Drug: Paclitaxel/cisplatin; Radiation: Intensity-modulated radiotherapy; Procedure: Esophagectomy

INTERVENTIONS:
Drug: Toripalimab — Patients received toripalimab 240 mg IVDRIP on days 1 and 22 during neoadjuvant radiotherapy.
  Other Names: JS-001
Drug: Paclitaxel/cisplatin — Patients received 4 cycles of paclitaxel/cisplatin (paclitaxel 50mg/m2 and cisplatin 25 mg/m2) on days 1, 8, 15, 22 during neoadjuvant radiotherapy.
  Other Names: TP
Radiation: Intensity-modulated radiotherapy — All patients received external-beam radiation using intensity-modulated radiotherapy. The prescribed dose is 44 Gy in 20 fractions over 4 weeks.
  Other Names: IMRT
Procedure: Esophagectomy — A transthoracic (Ivor-Lewis) esophagectomy is performed 6-8 weeks after CRT completion.

SUMMARY:
Neoadjuvant chemoradiotherapy (CRT) followed by surgery has become the standard treatment option for locally advanced esophageal cancer (EC). However, only 20% to 40% of EC patients can achieve pathologic complete response (pCR) after neoadjuvant CRT with favorable prognosis. Immunotherapy targeting the PD-1/PD-L1 checkpoints has demonstrated promising activity in advanced EC. The aim of this study was to evaluate the efficacy and safety of the combination of toripalimab (an anti-PD-1 antibody) combined with neoadjuvant CRT in locally advanced esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

1. A histopathological diagnosis of resectable thoracic esophageal squamous cell carcinoma with a pre-treatment clinical stage of T1-4aN1-3M0 or T3-4aN0M0 according to the 8th edition of the UICC staging system;
2. Patients who are anti-tumor treatment-naive;
3. Estimated life expectancy >6 months
4. Aged 18 to 70 years old of either gender
5. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥ 4.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L; b. platelets ≥ 100×109/L; c. hemoglobin ≥ 9g/dL; d. serum albumin ≥ 2.8g/dL; e. total bilirubin ≤ 1.5×ULN, ALT, AST and/or AKP ≤ 2.5×ULN; f. serum creatinine ≤ 1.5×ULN or creatinine clearance rate >60 mL/min;
6. PS score of 0-1;
7. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Patients who have been treated previously with anti-tumor therapy (including chemotherapy, radiotherapy, surgery, immunotherapy, etc.);
2. Known or suspected allergy or hypersensitivity to monoclonal antibodies, any ingredients of Toripalimab, and the chemotherapeutic drugs paclitaxel or cisplatin;
3. Patients who have a preexisting or coexisting bleeding disorder;
4. Other uncontrollable inoperable patients;
5. Female patients who are pregnant or lactating;
6. Inability to provide informed consent due to psychological, familial, social and other factors;
7. Presence of CTC grade ≥ 3 peripheral neuropathy;
8. A history of malignancies other than esophageal cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer
9. A history of diabetes for more than 10 years and poorly controlled blood glucose levels;
10. Patients who cannot tolerate chemoradiotherapy or surgery due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia.
11. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
12. A history of interstitial lung disease or non-infectious pneumonia;
13. A history of active pulmonary tuberculosis infection within 1 year or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal anti-tuberculosis treatment;
14. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate | Three working days after surgery
  The rate of pathologic complete response rate after neoadjuvant chemoradiotherapy.

SECONDARY OUTCOMES:
2-year overall survival | From date of randomization until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 24 months
  The 2-year overall survival of the whole group
2-year disease-free survival | From date of surgery until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months.
  The 2-year disease-free survival of the whole group
Incidence of Treatment-related Adverse Events as Assessed by CTCAE v4.0 | From the enrollment to the date of surgery
  The neoadjuvant treatment-related adverse events
R0 resection rate | Three working days after surgery
  The R0 resection rate of esophagectomy
Perioperative complication rate | From date of surgery to 30 days later
  The perioperative complication rate of esophagectomy
Perioperative mortality | From date of surgery to 30 days later
  The perioperative mortality of esophagectomy

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Fu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078
- [Result] Fu J, Wang F, Dong LH, Zhang J, Deng CL, Wang XL, Xie XY, Zhang J, Deng RX, Zhang LB, Wu H, Feng H, Chen B, Song HF. Preclinical evaluation of the efficacy, pharmacokinetics and immunogenicity of JS-001, a programmed cell death protein-1 (PD-1) monoclonal antibody. Acta Pharmacol Sin. 2017 May;38(5):710-718. doi: 10.1038/aps.2016.161. Epub 2017 Mar 20. PMID 28317872
- [Result] Tang B, Yan X, Sheng X, Si L, Cui C, Kong Y, Mao L, Lian B, Bai X, Wang X, Li S, Zhou L, Yu J, Dai J, Wang K, Hu J, Dong L, Song H, Wu H, Feng H, Yao S, Chi Z, Guo J. Safety and clinical activity with an anti-PD-1 antibody JS001 in advanced melanoma or urologic cancer patients. J Hematol Oncol. 2019 Jan 14;12(1):7. doi: 10.1186/s13045-018-0693-2. PMID 30642373
- [Derived] Mai Z, Kongjia L, Wang X, Xie X, Pang L, Yang H, Wen J, Fu J. Impaired TGF-beta signaling via AHNAK family mutations elicits an esophageal cancer subtype with sensitivities to genotoxic therapy and immunotherapy. Cancer Immunol Immunother. 2024 Sep 5;73(11):225. doi: 10.1007/s00262-024-03798-z. PMID 39235488
- [Derived] Chen R, Liu Q, Li Q, Zhu Y, Zhao L, Liu S, Chen B, Liu M, Hu Y, Lin T, Li J, Chen J, Lv Y, Fu J, Xi M, Yang H. A phase II clinical trial of toripalimab combined with neoadjuvant chemoradiotherapy in locally advanced esophageal squamous cell carcinoma (NEOCRTEC1901). EClinicalMedicine. 2023 Jul 26;62:102118. doi: 10.1016/j.eclinm.2023.102118. eCollection 2023 Aug. PMID 37560259